CLINICAL TRIAL: NCT05151237
Title: Incidence of Perioperative Hypothermia and Associated Risk Factors in Adults
Brief Title: Incidence of Perioperative Hypothermia in Adults
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Other Study IDs: 09.2021.296
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2021-12

CONDITIONS: Hypothermia; Anesthesia; Hypothermia Following Anesthesia
Keywords: hypothermia; perioperative; intraoperative; postoperative
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Measurement of body temperature — The patients' body temperature will be measured pre-, intra- and post-operatively via an infrared thermometer.

SUMMARY:
Perioperative hypothermia is associated with many complications, including surgical site infections, delayed wound healing, coagulopathy, prolonged hospital and intensive care unit length of stay. Perioperative close monitoring of the body temperature is important, and this is recommended by many clinical practice guidelines. In this study the investigators aimed to detect the incidence of perioperative hypothermia in adult patients in the operating room, and to detect the possible associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Any elective operation
* ASA I-III physical status

Exclusion Criteria:

* Emergency operations
* ASA IV-V physical status
* Open heart surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients scheduled for any elective operation (except for open heart surgery) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Body temperature | Perioperative
  Body temperature of the patients will be measured via infrared termometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No